CLINICAL TRIAL: NCT04487184
Title: Effect of the Different Methods of Kinesiology Taping on the Muscle Contraction Performance of Fatigued Biceps Brachii
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taoyuan General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TYGH107038
Record Dates: First submitted 2020-07-15; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2018-12

CONDITIONS: Muscle Fatigue
Keywords: Kinesiology tape; Fatigue; Muscle contraction performance
MeSH Terms: conditions — Fatigue | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Facilitation (Active Comparator): From origin to insertion
  Interventions: Other: Kinesiology taping
- Relaxation (Experimental): From insertion to origin
  Interventions: Other: Kinesiology taping
- Cross (Placebo Comparator): Cross the muscle fiber
  Interventions: Other: Kinesiology taping
- Control (Sham Comparator): No tape
  Interventions: Other: Kinesiology taping

INTERVENTIONS:
Other: Kinesiology taping — Recently, kinesiology tape is a common intervention in clinic and sport. The tension caused by tape elasticity and attachment techniques affects the effects that kinesiology tape produces, such as pain relief, circulation increase, proprioception enhancement, and muscle contraction improvement.
  Other Names: Kinesio tape

SUMMARY:
Recently, kinesiology tape is a common intervention in clinic and sport. According to the theory mentioned by the founder (Dr. Kenzo Kase), the elasticity of kinesiology tape has different effects from different taping skill. For muscle and fascia, taping could promote or inhibit contraction of muscle. For skeletal system, the intervention could correct posture and improve movement pattern through limiting joint mobility. For swelling, it may increase circulation of lymph during acute stage. However, whether these theories are feasible are still controversial in most studies.

The differences between results may be related to the high heterogeneity of taping method and outcome measures. On the other hand, there are lack of studies with high quality. The differences of taping method and skill should be considered for investigating the effect of kinesiology tape. And the performance of muscle contraction should be assessed by accurate instruments.

DETAILED DESCRIPTION:
Double-blind and crossover study design will be used in this study. The taping method is divided into 4 types: Tradition (from origin to insertion), Cross, New (from insertion to origin) and Control (non-taping). The order of types will be assigned to subjects randomly. The 4 types of taping will be applied in 2 days that one week apart. Ultimate physical rehabilitation system (Pris RS, BTE, USA) will be used to access the differences of muscle strength and muscular endurance between different taping skills. The aims are to investigate the effect of the different method of kinesiology tape on performance of fatigued biceps brachii.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults aged 20 years or older

Exclusion Criteria:

* Those who were unable to follow verbal instructions, had open wounds, or were allergic to kinesiology tape were excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Maximal Isometric Contraction Strength | Pre and immediately post test
  Ultimate physical rehabilitation system (Pris RS, BTE, USA) will be used to access the outcome
Change from Baseline Peak Contraction Speed | Pre and immediately post test
  Ultimate physical rehabilitation system (Pris RS, BTE, USA) will be used to access the outcome
Change from Baseline Maximal 10-s Power | Pre and immediately post test
  Ultimate physical rehabilitation system (Pris RS, BTE, USA) will be used to access the outcome
Change from Baseline Isokinetic Contraction Work | Pre and immediately post test
  Ultimate physical rehabilitation system (Pris RS, BTE, USA) will be used to access the outcome

CONTACTS AND LOCATIONS:
Overall Officials: Wu Ruo-Yan, Principal Investigator — Taoyuan General Hospital
Locations (1):
- Taoyuan General Hospital, Ministry of Health and Welfare, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
The datasets generated or analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Choi IR, Lee JH. Effect of kinesiology tape application direction on quadriceps strength. Medicine (Baltimore). 2018 Jun;97(24):e11038. doi: 10.1097/MD.0000000000011038. PMID 29901599